CLINICAL TRIAL: NCT04762160
Title: SYMPHONY-II: A Phase II Open-Label, Multicenter Trial of Oral Tazemetostat in Combination With Rituximab in Subjects With Relapsed/Refractory Follicular Lymphoma
Brief Title: SYMPHONY-2, A Trial to Examine Combination of Tazemetostat With Rituximab in Subjects With Relapsed/Refractory Follicular Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision to terminate EZH-1401 was solely due to company business decision.
Sponsor: Epizyme, Inc. (Industry)
Collaborators: Swedish Cancer Institute (Other)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZH-1401; NCT04590820 (obsolete NCT alias)
Record Dates: First submitted 2021-02-05; First posted 2021-02-21 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Follicular Lymphoma
Keywords: follicular lymphoma; relapse follicular lymphoma; refractory follicular lymphoma; rituximab; tazemetostat
MeSH Terms: conditions — Lymphoma, Follicular | interventions — tazemetostat; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tazmetostat in combination with rituximab (Experimental): Tazemetostat 800 mg BID is administered daily starting on Cycle 1 Day 1 (C1D1). Tazemetostat will be administered from C1D1 to the end of Cycle 24, for 24 months of therapy or until disease progression, unacceptable toxicity, or withdrawal of consent. Rituximab will be administered by either subcutaneous injection or IV infusion according to the regional product prescribing information, labeling and institutional guidelines. Rituximab will be administered at a dose of 375 mg/m2 on Day 1, 8, 15, and 22 of Cycle 1, and then on Day 1 of Cycles 3 through 6, accounting for an additional 4 doses, i.e., a total of 8 doses of rituximab in 6 cycles.
  Interventions: Drug: Tazemetostat; Combination Product: Rituximab

INTERVENTIONS:
Drug: Tazemetostat — Study Drug
  Other Names: EPZ-6438
Combination Product: Rituximab — Partner Drug
  Other Names: Rituximab Hyaluronidase

SUMMARY:
This study evaluates the safety and efficacy of combining the EZH2 inhibitor tazemetostat with rituximab in R/R FL subjects previously treated with at least 2 standard prior systemic treatment regimens where at least 1 anti-CD20-based regimen was used.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, open-label study of oral tazemetostat in combination with rituximab in subjects with relapsed or refractory (R/R) follicular lymphoma (FL). This study is designed to evaluate the safety and efficacy of tazemetostat in combination with rituximab in subjects previously treated with at least 2 standard prior systemic treatment regimens where at least 1 anti-CD20-based regimen was used, and used and features early futility stopping to maintain subject safety.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of 18 years of age and older
2. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol
3. Eastern Cooperative Oncology Group (ECOG) score of 0 </=, 1 or 2
4. Life expectancy (in the opinion of the investigator) of >3 months before enrollment
5. Have histologically confirmed FL, Grade 1 to 3a. Subjects may have R/R disease following at least 2 standard prior systemic treatment regimens where at least 1 anti- CD20-based regimen was used
6. Treatment recommended in accordance with the Groupe d'Etude des Lymphomes b Folliculaires (GELF) criteria
7. Meet the following laboratory parameters:

   1. Absolute neutrophil count (ANC) ≥ 750 cells/μL (0.75 x 109/L), or ≥ 500 cells/μL (0.50 x 109/L) in subjects with documented bone marrow involvement
   2. Platelet count ≥ 50,000 cells/μL (50 x 109/L), or ≥ 30,000 cells/μL (30 x 109/L) in subjects with documented bone marrow involvement, and without transfusion dependence
   3. Hemoglobin ≥ 8 g/dL
   4. Serum alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ Incl3.0 x ULN, unless related to disease involvement
   5. Total bilirubin ≤ 1.5 x ULN, unless due to disease involvement, Gilbert's syndrome, or hemolytic anemia
   6. Estimated creatinine clearance (ie, estimated glomerular filtration rate [eGFR] using Cockcroft-Gault) ≥ 40 mL/min
8. At least one bi-dimensionally measurable nodal lesion > 1.5 cm in its longest diameter by computed tomography (CT) scan or magnetic resonance imaging (MRI)
9. Any clinically significant toxicity related to a prior anticancer treatment (ie, chemotherapy, immunotherapy, and/or radiotherapy), except for alopecia, either resolved to ≤ Grade 1 per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 or is clinically stable and no longer clinically significant
10. Negative serologic or polymerase chain reaction (PCR) test results for acute or chronic hepatitis B virus (HBV) infection
11. Negative test results for hepatitis C virus (HCV) and human immunodeficiency virus (HIV).
12. Females of childbearing potential (FCBP) must have a negative serum pregnancy test (beta-human chorionic gonadotropin [β-hCG] test with a minimum sensitivity of 25 mIU/mL or equivalent units of β-hCG) at screening and within 24 hours prior to the first dose of study drug.
13. FCBP must either practice complete abstinence or agree to use a highly effective method of contraception beginning at least 28 days prior to the first dose of study drug, during study treatment (including during dose interruptions), for 6 months after tazemetostat discontinuation, and for 12 months after rituximab discontinuation. .
14. Male subjects must have had a successful vasectomy (with medically confirmed azoospermia) OR must either practice complete abstinence or agree to use a latex or synthetic condom during sexual contact with a FCBP from the first dose of study drug, during study treatment (including during dose interruptions), and for 3 months after study drug discontinuation.

Exclusion Criteria:

1. Prior exposure to Tazemetostat or other inhibitor(s) of EZH2
2. Grade 2b, mixed histology, or transformed FL
3. Treatment with any of the following anticancer therapies within the timeframe of a specific treatment prior to first dose of study drug:

   1. Cytotoxic chemotherapy within 21 days
   2. Noncytotoxic chemotherapy (e.g. small molecule inhibitor) within 14 days
   3. Nitrosoureas within 6 weeks
   4. Prior immunotherapy within 4 weeks
   5. Radiotherapy- within 6 weeks from prior radioisotope therapy; within 12 weeks from 50% pelvic or total body irradiation
   6. Any investigational treatment within 4 weeks or at least 5 half lives, whichever is shorter
4. History of solid organ transplant
5. Major surgery within 4 weeks of the start of study treatment
6. Thrombocytopenia, neutropenia, or anemia of Grade > 3 (per CTCAE v5.0 criteria) or any prior history of myeloid malignancies, including MDS/AML or MPN
7. Prior history of T-LBL/T-ALL
8. Unwillingness to exclude grapefruit juice-containing products, Seville oranges, and grapefruits from the diet and/ or consumed within 1 week of the first dose of study drug
9. Subjects taking medications that are known strong cytochrome P450 (CYP)3A inhibitors and strong or moderate CYP3A inducers (including St. John's wort)
10. Any uncontrolled illness
11. History of clinically significant cardiovascular abnormalities
12. History of clinically significant gastrointestinal (GI) conditions
13. Other diagnosis of cancer that is likely to require treatment in the next 2 years
14. Females who are pregnant or lactating/breastfeeding
15. Received a live virus vaccination within 28 days of first dose of rituximab
16. Concurrent participation in a separate investigational therapeutic study
17. Psychiatric illness/social situations that would interfere with study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (20):
- United States (20):
  - Alabama Oncology, Birmingham, Alabama
  - Compassionate Cancer Care, Fountain Valley, California
  - USOR/Rocky Mountain Cancer Centers, Boulder, Colorado
  - USOR/ Illinois Cancer Specialists, Niles, Illinois
  - XCancer/ Northwest Oncology & Hematology, Rolling Meadows, Illinois
  - Revive/Oakland Medical Group, Farmington Hills, Michigan
  - Revive/Hematology Oncology Associates of Rockland, Sterling Heights, Michigan
  - USOR/ NY Oncology Hematology, Albany, New York
  - East Carolina University, Greenville, North Carolina
  - USOR/ Oncology & Hematology Care Clinical Trials, Cincinnati, Ohio
  - XCancer/Dayton Physicians Network, Kettering, Ohio
  - XCancer/Tennessee Cancer Specialists, Knoxville, Tennessee
  - USOR/ Texas Oncology, Austin, Texas
  - USOR/Texas Oncology, Dallas, Texas
  - USOR/ Texas Oncology, San Antonio, Texas
  - USOR/ Texas Oncology, Tyler, Texas
  - USOR/Texas Oncology, Weslaco, Texas
  - USOR/Virginia Cancer Specialists, Gainesville, Virginia
  - USOR/Oncology & Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2, open-label study was conducted in participants with relapsed/refractory follicular lymphoma who received oral tazemetostat in combination with rituximab. The study was terminated early due to business reasons prior to enrolling the target number of participants needed to achieve target power and was insufficient to produce statistically reliable results.
Pre-assignment Details: This study was to include a 28-day screening period, a 2-year (24-cycle) treatment period, and a follow-up period. In treatment period, participants were to be treated in 28-day cycles with tazemetostat in combination with rituximab through Cycle 6 then tazemetostat alone through Cycle 24, for 24 months of therapy or until disease progression, unacceptable toxicity, or withdrawal of consent. Overall 5 participants were enrolled in the study.
Groups:
- Tazmetostat in Combination With Rituximab: Participants were to receive tazemetostat 800 milligram (mg) twice daily (BID) starting on Cycle 1 Day 1 until the end of Cycle 24, for 24 months of therapy or until study termination. Participants were also to receive rituximab, administered by either as subcutaneous (SC) injection or intravenous (IV) infusion according to the regional product prescribing information, labeling, and institutional guidelines. Rituximab was to be administered at a dose of 375 mg per square meter (m^2) on Cycle 1 Days 1, 8, 15, and 22 and then on Day 1 of Cycles 3 through 6, accounting for an additional 4 doses (i.e., a total of 8 doses of rituximab in 6 cycles). Each cycle was 28 days.
Period: Overall Study
Arm/Group | Tazmetostat in Combination With Rituximab
Started | 5
Completed | 0
Not Completed | 5
Not completed — Study terminated early due to business reasons | 5

BASELINE CHARACTERISTICS:
Population: The Safety population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline safety evaluation, regardless of enhancer of zeste homolog 2 (EZH2) mutation status (mutant-type [MT] or wild-type [WT]).
Groups:
- Tazmetostat in Combination With Rituximab: Participants were to receive tazemetostat 800 mg BID starting on Cycle 1 Day 1 until the end of Cycle 24, for 24 months of therapy or until study termination. Participants were also to receive rituximab, administered by either as SC injection or IV infusion according to the regional product prescribing information, labeling, and institutional guidelines. Rituximab was to be administered at a dose of 375 mg/m^2 on Cycle 1 Days 1, 8, 15, and 22 and then on Day 1 of Cycles 3 through 6, accounting for an additional 4 doses (i.e., a total of 8 doses of rituximab in 6 cycles). Each cycle was 28 days.
Arm/Group | Tazmetostat in Combination With Rituximab
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5
  Black or African American | 0
  Asian | 0
  American Indian or Alaska Native | 0
  Native Hawaiian or other Pacific Islander | 0
  Other/Unknown | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with WT EZH2 status who achieved a complete response (CR) or partial response (PR) according to the 2014 Lugano Classification as assessed by investigator and blinded independent review committee (IRC). CR = complete metabolic response per positron emission tomography-computed tomography (PET-CT) based response or complete radiologic response per CT-based response. PR = partial metabolic response per PET-CT-based response or partial remission per CT-based response.
Time Frame: Planned to be assessed during Cycles 3, 6, 12, 18, and 24.
Population: The study was terminated early due to business reasons and only five participants were enrolled, of whom only three were evaluable. No summary statistics are available given the limited data from the small number of evaluable participants and individual participant data are also not presented to protect the privacy of the individuals.
Arm/Group | Tazmetostat in Combination With Rituximab
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from first dose of study drug to the time of the earliest date of CR or PR per the 2014 Lugano Classification or death, whichever occurred first, as assessed by an IRC. CR= complete metabolic response per PET-CT based response or complete radiologic response per CT-based response. PR= partial metabolic response per PET-CT-based response or partial remission per CT-based response.
Time Frame: Planned to be assessed from first dose of study drug to earliest date of disease progression or death as assessed up to 24 months by an IRC
Population: as for outcome 1
Arm/Group | Tazmetostat in Combination With Rituximab
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the earliest date of CR or PR per the 2014 Lugano Classification to documented progression or death, whichever comes first, as assessed by an IRC. CR= complete metabolic response per PET-CT based response or complete radiologic response per CT-based response. PR= partial metabolic response per PET-CT-based response or partial remission per CT-based response.
Time Frame: Planned to be assessed from earliest date of CR or PR to documented progression or death as assessed up to 24 months by an IRC
Population: as for outcome 1
Arm/Group | Tazmetostat in Combination With Rituximab
Number analyzed (Participants) | 0

4. Secondary Outcome: ORR in a Subset of Participants With MT EZH2
Description: ORR was assessed according to 2014 Lugano Classification, in the pooled group regardless of mutation status and in a subset of participants with MT EZH2.
Time Frame: Planned to be assessed at the following timepoints: Cycles 3, 6, 12, 18, and 24
Population: as for outcome 1
Arm/Group | Tazmetostat in Combination With Rituximab
Number analyzed (Participants) | 0

5. Secondary Outcome: ORR in Rituximab Refractory Participants
Description: ORR was assessed according to 2014 Lugano Classification, in rituximab refractory participants.
Time Frame: Planned to be assessed at the following timepoints: Cycle 3, Cycle 6, Cycle 12, Cycle 18, and Cycle 24.
Population: as for outcome 1
Arm/Group | Tazmetostat in Combination With Rituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were assessed from the date of first dose of study treatment (Day 1) until 30 days after discontinuation of study treatment (approximately 462 days).
Description: The Safety population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline safety evaluation, regardless of EZH2 mutation status (MT or WT).
Arm/Group | Tazmetostat in Combination With Rituximab
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tazmetostat in Combination With Rituximab (N=5)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (3)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tazmetostat in Combination With Rituximab (N=5)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Testicular oedema (Reproductive system and breast disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Brachial plexopathy (Nervous system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to business reasons prior to enrolling the target number of participants needed to achieve target power and was insufficient to produce statistically reliable results and was not due to any safety concerns. No summary statistics are available given the limited data from the small number of evaluable participants and individual participant data are also not presented to protect the privacy of the individuals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT04762160/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT04762160/SAP_001.pdf